CLINICAL TRIAL: NCT01686230
Title: Effect of Acupuncture in Patients With Stable Angina Pectoris: an Open Label, Randomized, Controlled,Multi-center Clinical Study
Brief Title: Acupuncture in Patients With Stable Angina Pectoris
Acronym: ASAP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chengdu University of Traditional Chinese Medicine (Other)
Collaborators: Hunan University of Traditional Chinese Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 2012CB518501-4
Record Dates: First submitted 2012-08-23; First posted 2012-09-17 (Estimated); Last update posted 2020-02-17 (Actual); Status verified 2020-02

CONDITIONS: Angina, Stable
Keywords: acupuncture; Angina; Stable Angina Pectoris
MeSH Terms: conditions — Angina, Stable; Angina Pectoris | interventions — Acupuncture Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- acupoints on specific meridian (Experimental): Acupuncture plus foundation treatment。 We Select specific acpupoints on the heart and pericardium meridian.
  Interventions: Other: acupuncture; Drug: Basic treatment
- acupoints on the other meridian (Active Comparator): Acupuncture plus foundation treatment。We choose the acupoints on the other meridian。
  Interventions: Other: acupuncture; Drug: Basic treatment
- sham acupoints (Sham Comparator): Acupuncture plus foundation treatment。We use sham acupoints。
  Interventions: Other: acupuncture; Drug: Basic treatment
- waiting-list (Other): wait for the treatment，Only basic treatment, We will not treat the participants until they complete all the observations.
  Interventions: Drug: Basic treatment

INTERVENTIONS:
Other: acupuncture — In each session, we treat bilaterally, 3 times a week and 2 days off a week, each patient in the acupuncture treatment groups will receive 12 sessions of acupuncture treatment over 4 weeks. The whole study period is 20 weeks including 4-week baseline period,4-week treatment period, and 12-week follow-up period. we will investigate at 0 day,4week,8week,12week,16week after randomization。
  Other Names: Electro-acupuncture，Massage
  Arms: acupoints on specific meridian; acupoints on the other meridian; sham acupoints
Drug: Basic treatment — Each group in the basic treatment，Foundation treatment including health education and basic drug therapy.
  We recommend lifestyle modification for all patients. Modifications include increasing exercise; limiting alcohol consumption; and weight loss; quit smorking etc.
  Basic medication： Aspirin: 100mg qd; Metoprolol：25mg bid; Ramipril:5mg qd; Atorvastatin:20mg qn.
  Other Names: health education ， basic drug therapy

SUMMARY:
This trail aims to evaluate the efficacy of acupoints on the specific meridian for chronic stable angina pectoris, compared with acupoints on the other meridian, sham acupoints and waiting-list. And to confirm the specificity of acupoints on meridian.

DETAILED DESCRIPTION:
The basis of acupuncture is the theory of meridians and acupoints. Meridian and collaterals internally pertain to viscera, and externally spread over the extremities. An acupoint is the place where the visceral qi and meridian qi distributed in. besides acupoints are the stimulus points and reactive points for acupuncture to treat the diseases. Selecting the acupoints on the specific meridian is the basic principle of acupuncture. Recently, as to the existence of specificity of acupoints on the meridian has been questioned by many researchers. This trial using chronic stable angina pectoris as a carrier, select the acupoints on the hand shao yin heart meridian and hand jue yin pericardium meridian to treat chronic stable angina pectoris. Compared with acupoints on the other meridian and non-acupoints ,aiming to evaluate the efficacy, furthermore ,to confirm the existence of the specificity of acupoints on meridian.

ELIGIBILITY:
Inclusion Criteria:

1.Meet the diagnostic criteria of ACC/AHA angina pectoris of coronary heart disease.

2.35 ≤ age ≤ 80 years of age, both male and female.

3.The onset of angina pectoris≥3 months, and the frequency of angina attack≥2 a week.

4.Patients signed the informed consent.

Exclusion Criteria:

1. age≤35 or age≥80
2. Pregnant women or women in lactation or women of child bearing potential plan to conceive in the recent six months.
3. Combined with cardiovascular, digestive, respiratory, urinary, blood, nervous, endocrine system, severe primary disease clinical failed to effectively control the disease.
4. Complicated with mental disorders.
5. allergic constitution or bleeding disorder.
6. Patients accompany with acute coronary syndrome (including acute myocardial infarction, unstable angina), severe arrhythmias ( severe atrioventricular block, ventricular tachycardia, heartbeat influence the flow dynamics in supraventricular tachycardia, heartbeat frequent premature beats especially premature ventricular contractions ), atrial fibrillation, primary cardiomyopathy, valvular heart disease.
7. The blood pressure and blood glucose fail to meet the treatment targets.
8. Cardiovascular disease who had been treated with acupuncture during the previous three months.
9. Currently participating in other clinical trials.

Ages: 35 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 404 (Actual)
Dates: Start 2012-07 (Actual); Primary Completion 2017-07 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
Number of angina attacks | 16 weeks after inclusion
  The frequency of angina attack during 4-week.

SECONDARY OUTCOMES:
The severity of angina ( VAS score) | 0 day,4, 8, 12, 16 weeks after inclusion
  The VAS score evaluation angina pain severity
The dosage of nitroglycerin | 0 day,4, 8, 12, 16 weeks after inclusion
Six minute walk test | 0 day and 4 weeks after inclusion
  Six minute walk test in the evaluation of exercise tolerance
Dynamic ECG Observation of the changes of ST-T | 0 day and 4 weeks after inclusion
  Dynamic electrocardiogram in six minute walk test to do
The Seattle Angina Questionnaire ( SAQ ) score | 0 day,4, 8, 12, 16 weeks after inclusion
self-rating anxiety scale | 0 day,4, 8, 16 weeks after inclusion
The incidence of cardiovascular episode during the 4 months | 4, 8, 12, 16 weeks after inclusion
  The incidence of cardiovascular episode during the 4 months(develop into unstable angina, acute myocardial infarction, death)
Self-rating Depression Scale | 0 day,4, 8, 16 weeks after inclusion

CONTACTS AND LOCATIONS:
Overall Officials: fan-rong liang, Professor, Study Chair — Chengdu University of Traditional Chinese Medicine
Locations (1):
- Chengdu University of Traditional Chinese Medicine, Chengdu, Sichuan, China

REFERENCES:
- [Derived] Zhao L, Li D, Zheng H, Chang X, Cui J, Wang R, Shi J, Fan H, Li Y, Sun X, Zhang F, Wu X, Liang F. Acupuncture as Adjunctive Therapy for Chronic Stable Angina: A Randomized Clinical Trial. JAMA Intern Med. 2019 Oct 1;179(10):1388-1397. doi: 10.1001/jamainternmed.2019.2407. PMID 31355870
- [Derived] Li D, Yang M, Zhao L, Zheng H, Li Y, Chang X, Cui J, Wang R, Shi J, Lv J, Leng J, Li J, Liang F. Acupuncture for chronic, stable angina pectoris and an investigation of the characteristics of acupoint specificity: study protocol for a multicenter randomized controlled trial. Trials. 2014 Feb 5;15:50. doi: 10.1186/1745-6215-15-50. PMID 24499445